CLINICAL TRIAL: NCT01343407
Title: A Two-Part, Multicenter, Randomized, Clinical Trial to Study the Effects of Multiple Doses of MK-1029 on the Late Asthmatic Response to Lung Allergen Challenge in Asthmatics
Brief Title: A Two-part Study of the Effects of MK-1029 in Allergen-Challenged Asthmatics (MK-1029-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1029-003; 2010-022391-31 (EudraCT Number); MK-1029-003 (Other: Merck Protocol Number)
Record Dates: First submitted 2011-04-26; First posted 2011-04-28 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- MK-1029 60 mg (Experimental): Part 2 - Participants will receive 5 days of double-blind, once-daily MK-1029 60 mg followed by a 21-day washout in Period 2, 3, or 4 in a crossover design
  Interventions: Drug: MK-1029 10 mg; Drug: Placebo for MK-1029 10 mg
- MK-1029 500 mg (Experimental): Part 2 - Participants will receive 5 days of double-blind, once-daily MK-1029 60 mg followed by a 21-day washout in Period 2, 3, or 4 in a crossover design
  Interventions: Drug: MK-1029 100 mg; Drug: Placebo for MK-1029 100 mg
- Placebo (Placebo Comparator): Part II - Participants will receive 5 days of double-blind, once-daily MK-1029 60 mg followed by a 21-day washout in Period 2, 3, or 4 in a crossover design
  Interventions: Drug: Placebo for MK-1029 10 mg; Drug: Placebo for MK-1029 100 mg

INTERVENTIONS:
Drug: MK-1029 10 mg — Six capsules once daily for 5 days in Period 2, 3, or 4 in a crossover design
  Arms: MK-1029 60 mg
Drug: MK-1029 100 mg — Five capsules once daily for 5 days in Period 2, 3, or 4 in a crossover design
  Arms: MK-1029 500 mg
Drug: Placebo for MK-1029 10 mg — Six capsules once daily for 5 days in Period 1, and the same in Period 2, 3, or 4 in a crossover design."
  Arms: MK-1029 60 mg; Placebo
Drug: Placebo for MK-1029 100 mg — Five capsules once daily for 5 days in Period 2, 3, or 4 in a crossover design
  Arms: MK-1029 500 mg; Placebo

SUMMARY:
This was a 2-part study in participants with allergen-induced asthma. It included a procedural pilot component (Part 1). Part 1 tested the key procedures and timing of Part 2; no study drug was administered during Part 1. Part 2 included a pre-randomization placebo run-in (Period 1) and 3 treatment periods (Periods 2, 3, and 4) during which participants were randomized to receive double-blind placebo, MK-1029 60 mg or MK-1029 500 mg in a crossover design. The treatment periods were followed by a minimum 21-day washout. Part 2 assessed allergen-induced sputum eosinophils and allergen-induced late asthmatic response (LAR) compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

Parts 1 and 2

* Is male or a female of non-childbearing potential
* Has a history of allergen-induced asthma for at least 6 months
* Is judged to be in good health (other than asthma)
* Is able to perform reproducible pulmonary function testing
* Has a positive methacholine challenge test on Day -1
* Has an allergic response to house dust mite allergen as defined by positive skin prick test
* Is a nonsmoker and/ or has not used nicotine or nicotine-containing products for at least 12 months
* Has body mass index (BMI) ≥17 kg/m^2, but ≤33 kg/m^2

Part 2 only

* Must demonstrate a dual airway response to an allergen challenge in Period 1, decrease in FEV1 of at least 20% 0 to 2 hours after allergen challenge for early asthmatic response (EAR) and a positive late asthmatic response (LAR) to an inhaled allergen challenge as defined by a bronchoconstrictive response of at least 15% reduction in FEV1 3 to 8 hours after allergen challenge
* Can tolerate sputum induction and produce adequate sputum

Exclusion Criteria:

Parts 1 and 2

* Has a history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses additional risk to the participant
* Has recent (4 weeks) or ongoing upper or lower respiratory tract infection
* Is unable to refrain from or anticipates the use of any medication other than the ones permitted in this study
* Has taken oral, intramuscular, intra-articular, high-potency topical or orally inhaled corticosteroids within 8 weeks
* Has taken the following medications outside the washout margins: nasal corticosteroids and anti-leukotrienes within 3 weeks; inhaled long-acting β2-agonists, long-acting antihistamines (e.g., loratadine, sustained-release agents), intra-nasal anticholinergics over-the-counter decongestants within 1 week; short-acting oral decongestants, short-acting antihistamines (e.g., chlorpheniramine) within 48 hours
* Consumes excessive amounts of alcohol or caffeinated beverages
* Has had major surgery, donated or lost 1 unit of blood or participated in another investigational study within 3 months
* Has a history of severe allergies, or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Is a nursing mother
* Has a history of receiving anti-immunoglobulin E (IgE) or immunotherapy
* Has a history of serious allergies to drugs or a history of hypersensitivity to mometasone furoate or any of its inactive ingredients such as lactose, or inhaled salbutamol, antihistamines, or any

other potential asthma/anaphylaxis rescue medication

Part 2 only

- Has a decline in FEV1 of 70% or greater from the post allergen diluent baseline and/or FEV1 <1.0L or has symptomatic drop in FEV1 associated with shortness of breath unresolved with bronchodilators within a reasonable timeframe (60 minutes) after the allergen challenge study in Period 1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-04-19 (Actual); Primary Completion 2012-01-09 (Actual); Study Completion 2012-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a 2-part study. Part 1 was a procedural pilot, performed first and including placebo run-in (Period 1), with no study drug administration. Part 2 began with pre-randomization placebo run-in (Period 1), followed by 3 randomized, crossover treatment periods (Periods 2, 3, and 4). The Participant Flow applies only to randomized participants.
Groups:
- Sequence 1: Placebo→MK-1029 60 mg→ MK-1029 500 mg. Participants received 5 days of crossover treatment (once-daily dosing) in 3 periods, followed by a minimum 21-day washout between treatment periods.
- Sequence 2: MK-1029 60 mg→MK-1029 500 mg→Placebo. Participants received 5 days of crossover treatment (once-daily dosing) in 3 periods, followed by a minimum 21-day washout between treatment periods.
- Sequence 3: MK-1029 500 mg→Placebo→ MK-1029 60 mg. Participants received 5 days of crossover treatment (once-daily dosing) in 3 periods, followed by a minimum 21-day washout between treatment periods.
- Sequence 4: Placebo→MK-1029 500 mg→ MK-1029 60 mg. Participants received 5 days of crossover treatment (once-daily dosing) in 3 periods, followed by a minimum 21-day washout between treatment periods.
- Sequence 5: MK-1029 500 mg→MK-1029 60 mg→Placebo. Participants received 5 days of crossover treatment (once-daily dosing) in 3 periods, followed by a minimum 21-day washout between treatment periods.
- Sequence 6: MK-1029 60 mg→Placebo→ MK-1029 500 mg. Participants received 5 days of crossover treatment (once-daily dosing) in 3 periods, followed by a minimum 21-day washout between treatment periods.
Period: First Treatment Period (Part 2)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started (Allergen challenge was done 1 hour after dosing on Day 5 of each treatment period.) | 2 | 2 | 3 | 3 | 3 | 3
Completed | 2 | 2 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: First Washout (Part 2)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 2 | 2 | 3 | 3 | 3 | 3
Completed | 2 | 2 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Treatment Period (Part 2)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started (Allergen challenge was done 1 hour after dosing on Day 5 of each treatment period.) | 2 | 2 | 3 | 3 | 3 | 3
Completed | 2 | 2 | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Period: Second Washout (Part 2)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 2 | 2 | 2 | 3 | 3 | 3
Completed | 2 | 2 | 1 | 3 | 3 | 3
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Period: Third Treatment Period (Part 2)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started (Allergen challenge was done 1 hour after dosing on Day 5 of each treatment period.) | 2 | 2 | 1 | 3 | 3 | 3
Completed | 2 | 2 | 1 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomized Participants: Crossover treatment with MK-1029 60 mg, MK-1029 500 mg, and matching placebo
Arm/Group | Randomized Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Percent (%) Eosinophils in Induced Sputum At 8 Hours Post Allergen
Description: The effect of MK-1029 on the reduction of percent (%) sputum eosinophils following allergen challenge with standardized cat pelt or hair (CPH) allergen extract was assessed. Baseline % eosinophils were measured before treatment (and pre-allergen challenge) on Day -1. The change from baseline in allergen-induced % sputum eosinophils at 8 hr post allergen challenge testing on Day 5 was analyzed using a repeated measures linear mixed effects model with treatment, period, time, time-by-treatment interaction as fixed factors, and participant as a random factor. Outcome Measure 6 shows % eosinophil values at baseline.
Time Frame: Baseline (Day -1) and Day 5 (8 hours after allergen challenge in each treatment period)
Population: Participants who comply with the protocol sufficiently to ensure data obtained will be likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Groups:
- MK-1029 60 mg: Participants received 5 days of treatment with MK-1029 60 mg (once-daily dosing) in 3 periods, followed by a minimum 21-day washout between treatment periods
- MK-1029 500 mg: Participants received 5 days of treatment with MK-1029 500 mg (once-daily dosing) in 3 periods, followed by a minimum 21-day washout between treatment periods
- Placebo: Participants received 5 days of treatment with placebo (once-daily dosing) in 3 periods, followed by a minimum 21-day washout between treatment periods
Arm/Group | MK-1029 60 mg | MK-1029 500 mg | Placebo
Number analyzed (Participants) | 11 | 12 | 9
Percent change | -10.6 [-22.5 to 1.3] | -7.3 [-18.3 to 3.6] | 11.6 [-1.0 to 24.3]
Statistical Analysis 1: Comparison: MK-1029 60 mg vs Placebo; Test type: Other; p = 0.011, Linear mixed effects model; Difference in Least Squares Means (LSM) = -22.2, 90% CI 2-sided [-35.7 to -8.7]
Statistical Analysis 2: Comparison: MK-1029 500 mg vs Placebo; Test type: Other; p = 0.023, Linear mixed effects model; Difference in LSM = -18.9, 90% CI 2-sided [-32.1 to -5.8]

2. Primary Outcome: Forced Expiratory Volume in One Second (FEV1) From 3 to 8 Hours Postdose (AUC3-8hr) During the Late Asthmatic Response (LAR)
Description: The effect of MK-1029 on the FEV1 AUC(3-8hr) during LAR was assessed. The unit of measure for an FEV1 AUC value is L*hr. The effect of treatment on LAR was assessed as the percent-fall in FEV1 AUC(3-8hr), evaluated by spirometry following allergen challenge on Day 5. The FEV1 AUC(3-8hr) during LAR was analyzed using a linear mixed effects model with treatment and period as fixed factors and participant as a random factor.
Time Frame: From 3 to 8 hours after allergen challenge on Day 5 of each treatment period
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: L*hr
Arm/Group | MK-1029 60 mg | MK-1029 500 mg | Placebo
Number analyzed (Participants) | 14 | 16 | 15
L*hr | 41.24 [18.16 to 93.66] | 49.76 [31.02 to 79.83] | 86.37 [55.79 to 133.70]
Statistical Analysis 1: Comparison: MK-1029 60 mg vs Placebo; Test type: Other; p = 0.006, Linear mixed effects model; LS Mean Ratio (LSMR) = 0.48, 90% CI 2-sided [0.32 to 0.72]; % Inhibition: 52.2 (90% CI: 28.3, 68.2). The % Inhibition of FEV1*hr (reduction of the allergen-induced LAR) for MK-1029 vs Placebo was calculated as 100*(1-LSMR)
Statistical Analysis 2: Comparison: MK-1029 500 mg vs Placebo; Test type: Other; p = 0.012, Linear mixed effects model; LS Mean Ratio (LSMR) = 0.58, 90% CI 2-sided [0.41 to 0.81]; % Inhibition: 42.4 (90% CI: 19.3, 58.8) The % Inhibition of FEV1*hr (reduction of the allergen-induced LAR) for MK-1029 vs Placebo was calculated as 100*(1-LSMR)

3. Secondary Outcome: Percent Inhibition of the Expression of Cluster of Differentiation (CD)11b on Blood Eosinophils
Description: The concentration of CD11b in whole blood samples was assessed. The percent-inhibition of CD11b (a cell-surface biomarker on activated eosinophils) was assessed following inhaled allergen challenge on Day 5. Inhibition of CD11b expression was assessed by analyzing the % inhibition of CD11b expression from baseline (Day -1) using a linear mixed-effects model with period, treatment, time, and treatment by time as fixed terms and subject as a random term. Outcome Measure 7 shows CD11b expression values at baseline.
Time Frame: Baseline (Day -1, predose), 24 hours after allergen challenge on Day 5 in each treatment period
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of inhibition
Arm/Group | MK-1029 60 mg | MK-1029 500 mg | Placebo
Number analyzed (Participants) | 13 | 16 | 15
Percentage of inhibition | 89.9 [71.8 to 108.0] | 87.4 [71.2 to 103.5] | 4.1 [-12.6 to 20.8]
Statistical Analysis 1: Comparison: MK-1029 60 mg vs Placebo; Test type: Other; p < 0.001, Linear mixed effects model; LSM Difference = 85.84, 90% CI 2-sided [65.3 to 106.4] — Full inhibition is ≥74% inhibition of blood eosinophil CD11b expression at trough
Statistical Analysis 2: Comparison: MK-1029 500 mg vs Placebo; Test type: Other; p < 0.001, Linear mixed effects model; LSM Difference = 83.29, 90% CI 2-sided [63.9 to 102.7] — Full inhibition is ≥74% inhibition of blood eosinophil CD11b expression at trough

4. Primary Outcome: Number of Participants With an Adverse Event (AE)
Description: The number of participants who had at least one adverse event (AE) during study treatment and follow-up was assessed. An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product.
Time Frame: Up to 26 days in each treatment period
Population: All randomized participants who received at least one dose of study treatment and had follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1029 60 mg | MK-1029 500 mg | Placebo
Number analyzed (Participants) | 14 | 16 | 16
Participants | 11 | 10 | 11

5. Primary Outcome: Number of Participants Discontinuing Treatment Due to an AE
Description: The number of participants who discontinued study treatment due to an AE was assessed. An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product.
Time Frame: Up to 5 days in each treatment period
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1029 60 mg | MK-1029 500 mg | Placebo
Number analyzed (Participants) | 14 | 16 | 16
Participants | 0 | 0 | 1

6. Other Pre Specified Outcome: Baseline (Pre-Treatment) Percent (%) Eosinophils
Description: Baseline values of the percent (%) sputum eosinophils were measured pre-antigen challenge on Day -1. The baseline % eosinophil values were provided to assess the change from baseline after treatment.
Time Frame: Baseline (Day -1), pre-antigen challenge
Population: Participants who were compliant with the protocol sufficiently to ensure their data would be likely to exhibit the effects of treatment were included.
Measure: Mean (Full Range); unit: % sputum eosinophils
Arm/Group | MK-1029 60 mg | MK-1029 500 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 12
% sputum eosinophils | 18.42 [0.47 to 80.56] | 17.04 [0.66 to 78.22] | 11.99 [0.48 to 23.40]

7. Other Pre Specified Outcome: Baseline Expression of Cluster of Differentiation (CD)11b on Blood Eosinophils
Description: Baseline values for the antibody-specific expression of CD11b in whole blood samples, as obtained by flow cytometry, were obtained. The baseline CD11b values were obtained before treatment with MK-1029 60 mg, MK-1029 500 mg, or placebo, and were used to assess the effects of treatment.
Time Frame: Day 1, predose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Antibody fluorescence units
Arm/Group | MK-1029 60 mg | MK-1029 500 mg | Placebo
Number analyzed (Participants) | 13 | 16 | 15
Antibody fluorescence units | 62619 (28790) | 62254 (13690) | 63398 (22022)

ADVERSE EVENTS:
Time Frame: Up to 26 days in each treatment period
Description: One participant had an episode of respiratory distress (a serious AE) during the placebo run-in, and was not randomized to study treatment. The at-risk population for AEs is all participants who received study drug in a treatment period.
Groups:
- 60 mg MK-1029: Participants received 5 days of treatment with MK-1029 60 mg (once-daily dosing) in 3 periods, followed by a minimum 21-day washout between treatment periods
- 500 mg MK-1029: Participants received 5 days of treatment with MK-1029 500 mg (once-daily dosing) in 3 periods, followed by a minimum 21-day washout between treatment periods
Arm/Group | 60 mg MK-1029 | 500 mg MK-1029 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 11/14 | 10/16 | 11/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 60 mg MK-1029 (N=14) | 500 mg MK-1029 (N=16) | Placebo (N=16)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 3 (3) | 0 (0) | 3 (6)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 6 (7) | 5 (7)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 6 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This study is intended for publication, even if terminated prematurely. The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines.